CLINICAL TRIAL: NCT04000191
Title: Numb the Bum: Ice as an Adjunct for Local Anesthesia During Anorectal Surgeries
Brief Title: Ice as an Adjunct for Local Anesthesia During Anorectal Surgeries
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was neer started and PI left the institution.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-38798
Record Dates: First submitted 2019-06-17; First posted 2019-06-27 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia, Local
Keywords: ice; elective anorectal surgery; anesthesia care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Usual monitored anesthesia care (MAC) (Active Comparator): Monitored anesthesia care (MAC) administered by anesthesiology and injection of local anesthesia by the operating surgeon.
  Interventions: Procedure: MAC
- MAC and perianal ice (Experimental): Monitored anesthesia care (MAC) administered by anesthesiology, application of ice to the perianal area after it is prepared with betadine, and injection of local anesthesia by the operating surgeon.
  Interventions: Procedure: MAC; Other: Perianal ice application

INTERVENTIONS:
Procedure: MAC — Monitored anesthesia care (MAC) administered by anesthesiology and Injection of local anesthesia mixture of 1% lidocaine with epinephrine and 0.25% Marcaine by the operating surgeon.
Other: Perianal ice application — Application of ice to the perianal area after the area is prepared with betadine, prior to injection of local anesthesia by the surgeon.
  Arms: MAC and perianal ice

SUMMARY:
The purpose of this study is to determine, among patients receiving elective anorectal surgery, does application of ice to the perianal area prior to the procedure, lead to use of decreased amounts of intravenous (IV) anesthesia? Anorectal surgeries for hemorrhoids, fistulas and fissures are done on an outpatient basis under monitored anesthesia care. This means patients get sedating medications through an IV but often do not require intubation. The difficulty with monitored anesthesia is balancing patient comfort against the risk of apnea (not breathing due to over sedation). Application of ice to the perianal area may help increase patient comfort, decrease the amounts of medications given for sedation and therefore decrease risk and increase recovery from the anesthesia.

DETAILED DESCRIPTION:
The study design will be a randomized control trial of adults undergoing elective surgery for hemorrhoids, fistulas, perianal/perirectal abscess and anal fissure. Participants will be randomized in a 1 to 1 ratio using a random number generator to two arms to the study - usual care vs. usual care plus ice to numb the anal area prior to incision.

The outcomes will be measured the same day as the surgery. Prior to leaving the operating room the anesthesia team will share with the surgeon the amount of each drug they administered. A comfort score will be recorded by the study personnel in the recovery area prior to discharge for each participant.

ELIGIBILITY:
Inclusion Criteria:

-Patient with planned minor elective colorectal surgery (eg for hemorrhoids, perianal abscess, fistula in ano, anal fissure, pilonidal cysts, or anal condyloma)

Exclusion Criteria:

-Patient who requires general anesthesia as part of the initial anesthesia plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Amount of drugs administered to each participant | Within 1 days after each surgical procedure
  The total number of milligrams for each medication administered by the anesthesiologist will be recorded (eg Versed, Fentanyl, Propofol, etc)

SECONDARY OUTCOMES:
Participant self pain assessment in the recovery area | Within 2 hours after each surgical procedure
  A validated instrument that consists of a 10cm line will be used to assess post-operative discomfort. Each participant will be asked to make a mark on the line to indicate their level of pain. The left end of the line indicates a score of "No Pain" and the right end of the line indicates "Worst Pain." The location of the mark will be measured and the pain score will be a ratio of the distance of the mark measured from the "No Pain" end over the total length of the line (10cm).

CONTACTS AND LOCATIONS:
Overall Officials: Uma R Phatak, MD MS, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No